CLINICAL TRIAL: NCT02622308
Title: The Effects of Intermittent Negative Pressure on Peripheral Circulation in Dialysis Patients and Patients With Lower Limb Ischemia and Leg Ulcers
Brief Title: The Effects of INP on Peripheral Circulation in Dialysis Patients and Patients With PAD and Leg Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of recruitment
Sponsor: Oslo University Hospital (Other)
Collaborators: Otivio AS (Industry); University of Oslo (Other)
Responsible Party: Principal Investigator, Jonny Hisdal, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1318
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-08

CONDITIONS: Renal Disease; Peripheral Arterial Disease; Arterial Leg Ulcers
Keywords: Arterial leg ulcers; Intermittent Negative Pressure; Peripheral Circulation; Wound healing; Peripheral blood flow
MeSH Terms: conditions — Kidney Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-case design (Experimental): The study design will be a non-randomized clinical trial with single-subject baseline design (also called single-case baseline design) where each patients act as their own controls:
  Observations (A) will be taken before and after a 8-week intervention period. We plan to introduce a 4-week INP-treatment period ('FlowOx™) (B) using the same outcome variables that were used as baseline measures. If the patient demonstrates improvements in outcome variables after the first treatment period (B1), the patient will be asked to continue INP therapy for another 4-week period, before a final assessment after a total of 8-week intervention period (B2) (A-B-B design).
  Interventions: Device: FlowOx™

INTERVENTIONS:
Device: FlowOx™ — FlowOx™ uses intermittent negative and atmospheric pressure, and is intended for use as an adjunct non-invasive therapy for the treatment of reduced peripheral circulation. Negative pressure cycles are created by alternating between removing air and venting the vacuum-chamber to atmospheric pressure. The vacuum cycle is controlled by the Control Unit (Pump). FlowOx™ is designed to assists wound healing indirectly by improving blood flow to the affected limb and augmenting the wound healing effect of the contact dressings and any associated medication. Treatment is planned to be applied while the participants are seated and it does not interfere with other activities normally enjoyed while seated. Treatment is recommended for one to two hours per session aiming to improve blood flow in the affected area and thus the clinical outcomes.
  Other Names: Intermittent negative pressure device

SUMMARY:
This experimental study will look at the effects of INP therapy for two patient groups: 1) patients with reduced peripheral circulation and chronic wounds in patients with renal disease (dialysis patients); 2) and peripheral arterial disease and leg ulcers. The project is designed as a non-randomized clinical trial with single-subject multiple baseline design. Also the intervention will be subjected on the same leg for each individual throughout the study period. The other leg will act as a control. A baseline measure with patient history collection will be performed before a four-week intervention period. These measures include: Segmental pulse-volume-recording, Segmental skin perfusion pressure with a laser Doppler sensor and a pressure cuff to evaluate reactive hyperemia (Sensilase, Väsamed) and a health survey (SF-12/EQ-5D-5L) or similar. After four weeks and eight weeks of intervention, the same tests will be repeated. A final follow-up test will be two weeks after cessation of the intermittent negative pressure intervention. The study will look at the effect of INP on renal failure patients who are given dialysis at a dialysis center located at Oslo University Hospital, Ullevål. Otivio AS has supplied the FlowOx devices and provided the necessary training to perform this project. Outcome variables assessed before, during and after the 10-week study period will be: wound healing, quality of life, skin perfusion pressure and segmental pulse-volume recording. The aim of this project is to prospectively examine and elucidate the effect of intermittent negative pressure therapy on clinically relevant measures related to the reduction of peripheral macro- and microcirculation in patients with renal failure undergoing dialysis treatment.

The hypothesis of the study is:

* Application of INP in patients with renal failure, by the use of the FlowOx™ device, will improve wound healing and peripheral circulation in the foot compared to before treatment (baseline) in patients undergoing dialysis treatment.
* Application of INP in patients with PAD, by the use of the FlowOx™ device, will improve macro- and microcirculation and wound healing in the foot compared to before treatment (baseline) in patients with chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Age: 18-96 years
* Affected foot/shoe size <46 (approximate foot length< 29,5 cm)
* Receiving hemodialysis ≥3 times per week for 1 hour per treatment OR
* Peripheral arterial disease and leg ulcer

Exclusion criteria:

* Incapable to consent voluntarily, i.e. patients who are not able to consent due to their mental status, or who are not willing or able to perform the negative pressure therapy in a sitting position
* Not adhering to the INP therapy program
* Patients with an expected life-span less than 3 months
* Patients in whom the remaining limb is non-functional, for example due to previous stroke
* Patients in which a deep venous thrombosis or pulmonary embolism is suspected
* Limbs with uncontrolled infection
* Previous lumbar sympathectomy
* Bilateral amputation of lower extremity

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
Segmental Skin Perfusion Pressure | 8 weeks
  Fully automated and quantitative evaluation of microcirculatory perfusion in the skin of the foot and leg (Sensilase, Vasamed, USA).
  Multiple levels can be assessed on limbs; bilateral measurement helps to manage test time Not susceptible to interference effects from medial calcification Requires use of pressure cuffs to occlude blood flow for specified time period in order to evaluate reactive hyperemic response to controlled release of pressure Graphical output of pressure and perfusion during cuff deflation indicates the pressure (mmHg) at which skin perfusion is found to return in addition to pressure contour
Life Quality (SF-12 or EQ-5D-5L) | 8 weeks
  SF-12 or EQ-5D-5L
Pulse Volume Recording / segmental volume plethysmography (PVR) | 8 weeks
  PVR shows variations in the volume of blood passing through a limb during each cardiac cycle. The instrument that will be used to measure PVR for this study is Sensilase (Vasamed, USA) OR MacroLab (STR Teknikk, strteknikk.no, Aalesund, Norway).
  Multiple levels can be assessed on limbs. The measures are not susceptible to interference effects from medial calcification.
Wound healing (Measuring wound diameter and length) | 8 weeks
  Measurement of healing to provide a means by which progress over time to wound closure can be identified. A wound nurse will take pictures at study start and at follow-up.
Ankle-Brachial Pressure Index (ABPI) | 8 weeks
  The ratio of the blood pressure at the ankle (dorsal pedis artery/posterior tibial artery) to the blood pressure in the upper arm (brachial artery)

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Hisdal, PhD, Principal Investigator — Oslo University Hospital - Aker
Locations (1):
- Oslo University Hospital - Ullevål, Department of Nephrology, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided